CLINICAL TRIAL: NCT04456257
Title: The Efficacy of 1,064-nm Picosecond Laser With Microlens Array for the Treatment of Abdominal Striae Distensae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si 591/2561
Record Dates: First submitted 2020-05-26; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Striae Alba
Keywords: striae alba, fractional picosecond laser, stretch marks
MeSH Terms: conditions — Striae Distensae | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fractional Picosecond 1,064 nm laser (Experimental): The subjects with abdominal striae alba were treated with a fractional picosecond 1,064 nm laser
  Interventions: Device: fractional picosecond 1,064 nm laser

INTERVENTIONS:
Device: fractional picosecond 1,064 nm laser — The parameter of laser was 8-mm spot size, 0.6 mJ/cm2, 750 ps, 10 Hz, 2 passes. The treatment was done in every 4 weeks for 4 sessions.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of a fractional 1,064 nm picosecond laser for the treatment of striae alba.

DETAILED DESCRIPTION:
Striae distensae are atrophic dermal scars that can cause psychosocial distress on affected patients. Despite numerous available therapeutic modalities, no gold standard therapy has been established. Picosecond lasers are a newer advancement in lasers that have primarily used in the treatment of tattoos. A fractional 1064-nm picosecond laser has recently become available for the treatment of pigmentation and skin rejuvenation. The main mechanism of action is tissue ablation via laser induced optical breakdown (LIOB) which occur when pulse intensity is high enough to strip electrons and generating plasma, the plasma absorbs the remaining laser energy forming a cavitation bubble within the dermis which has been demonstrated to improve fine wrinkles and acne scar through the stimulation of collagen formation.

ELIGIBILITY:
Inclusion Criteria:

* Striae alba on abdomen for more than 3 months
* Fitzpatrick skin type III-V

Exclusion Criteria:

* Pregnancy and breastfeeding
* Previous topical treatment, filler injection, chemical peel or laser treatment within 6 months before starting the study
* History of using Isotretinoin
* Photosensitive dermatoses, Infection, eczema
* Past history or family history of malignancy
* History of herpes infection
* History of hypertrophic scar or keloid, connective tissue disease
* History of collagen or elastin disease
* History of smoking
* Significant fluctuations in weight in the past 6 months

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in striae roughness by Antera 3D image | change from baseline in striae roughness score at 6 months
Change in average Melanin index by Antera 3D image | change from baseline in average melanin index at 6 months
Change in melanin variation index by Antera 3D image | change from baseline in melanin variation index at 6 months

SECONDARY OUTCOMES:
Investigator assessment scores | Baseline, 1, 3 and 6 months after final treatment
  Clinical improvement was evaluated by comparing pre and post photographs by 2 independent investigators.
Patient satisfaction scores | Baseline, 1, 3, and 6 months after final treatment
  patient satisfaction questionnaire was done by grading on a scale of 0 to 4; 0: no improvement, 1: <25% improvement, 2: 25-50% improvement, 3: 51-75% improvement, 4: > 75% improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand